CLINICAL TRIAL: NCT03203174
Title: The Use of Microneedles With Topical Botulinum Toxin for Treatment of Palmar Hyperhidrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 561309
Record Dates: First submitted 2015-12-01; First posted 2017-06-29 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Hyperhidrosis
Keywords: microneedle; botulinum toxin; botox; palmar hyperhidrosis; sweating; hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subject's received treatment to one palm and the other palm was used as a control.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Split-hand Microneedle Botulinum Toxin A (Experimental): One palm with microneedle pretreatment prior to application of topical botulinum toxin A
  Interventions: Device: Microneedle; Drug: Botulinum Toxin Type A; Other: Saline
- Split-hand Sham Microneedle Botulinum Toxin A (Sham Comparator): Contralateral palm with sham microneedle pretreatment prior to application of topical botulinum toxin A
  Interventions: Device: Sham Microneedle; Drug: Botulinum Toxin Type A; Other: Saline

INTERVENTIONS:
Device: Microneedle — Microneedles are small needles used to create holes in the stratum corneum (top layer of skin) with relatively low amount of pain.
  Arms: Split-hand Microneedle Botulinum Toxin A
Device: Sham Microneedle — Flat roller with no needles on the roller
  Arms: Split-hand Sham Microneedle Botulinum Toxin A
Drug: Botulinum Toxin Type A — Botulinum toxin type A will be applied to the palm
Other: Saline — Saline applied to the palm

SUMMARY:
Hyperhidrosis or sweating of palms results from the overactivity of sweat glands and leads to psychosocial impairment with reduction in quality of life in those that are affected. Injection of botulinum toxin has been shown to be effective in reducing the symptoms of hyperhidrosis with associated improvement in quality of life, but is usually very painful. Microneedles are a different modality for transdermal drug penetration without the pain. This study aims to understand if botulinum toxin A can be delivered topically after microneedle pretreatment in hopes of developing a minimally painful treatment protocol for treatment of palmar hyperhidrosis.

DETAILED DESCRIPTION:
Split-hand Microneedle group: After the subject has been consented, the Treatment Visit will commence. Subjects will be randomized into one of two groups. Binary randomization for microneedle pretreatment of the right vs. the left hand (Dominant hand has higher strength which may skew side effect reporting of weakness).

The evaluation of sweat production will be done using the subjective patient reported Hyperhidrosis Disease Severity Scale (HDSS) and objective gravimetric measurement. Hyperhidrosis Disease Severity Scale (HDSS) is a scale from 1 to 4. Values of 1 or 2 represent Mild/moderate disease, and 3 or 4 represent severe disease. Successful treatment is indicated by improvement from 3 or 4 to 1 or 2. One point improvement in HDSS score is associated with 50% reduction in sweat production and a two-point improvement with an 80% reduction, according to the Canadian Hyperhidrosis Advisory Committee.

Gravimetric measurement includes collecting sweat secretion on standardized filter. Prior to any measurements, the subject will be asked to sit in a climate-controlled room for 15 min to allow for acclimatization. Filter paper is first weighed on a high-precision laboratory scale. The filter papers are then placed in the subject's palms for 5 minutes, and weighed again. This technique has already been used in other studies of hyperhidrosis [5]. The difference in the weight (g) will allow calculation of sweat secretion in grams per 5 minutes.

The subject's palm will be cleansed with gauze. Then the microneedle pretreatment versus sham microneedle pretreatment will be performed. This will consist of rolling the microneedles or sham microneedles into the skin for several seconds on the sides of the palm that have respectively been randomized to the microneedle or control treatment. Sham microneedles will consist of a flat roller without the presence of the microneedles. The microneedles are solid and are long enough to penetrate the stratum corneum and enter the epidermis. Microneedles that are less than 700 micrometers in length have been shown to induce minimal pain, and our ongoing work with microneedles that were 650 micrometers in length was rated a 1 out of 10 on a visual analog pain scale. For this study, subjects will rate pain on a visual analog scale after the microneedle pretreatment as well.

Next a Transepidermal Water Loss Meter (Tewameter) will be used to measure the water evaporation gradient on the skin. Measurements will be performed with non-invasive devices that have been widely used for the study of skin barrier function. Each device has a flat-top electrode (approximate diameter of 1cm) that will come in contact with the skin surface during measurements. This device does not deliver any energy into the skin. The subjects will not experience discomfort during and after the measurements. The electrode tip will be cleaned with alcohol wipes between subjects.

Next, the subject will asked to grade their discomfort with the pretreatment step on a 10 cm visual analog pain scale.

Next, botulinum toxin A solution will be mixed per standard protocol in the dermatology clinic and will be applied and evenly spread over the palm. This will be followed by occlusion with an occlusive wrap such as saran wrap or a silicone based gel. The subject will be asked to keep the saran wrap in place for 1 hour. Botulinum toxin A is an FDA approved product for the treatment of hyperhidrosis.

Follow-up visits will be at 4-6 weeks post treatment. During the follow-up visit the patient will be asked about side effects or any adverse events. Also a repeat evaluation of sweat production will be done using the subjective patient reported Hyperhidrosis Disease Severity Scale (HDSS) and objective gravimetric measurement. They will also complete a global satisfaction survey.

Split-hand Botulinum Toxin A group: After the subject has been consented, the Treatment Visit will commence. Subjects will be randomized into one of two groups. Binary randomization for botulinum toxin A of the right vs. the left hand (Dominant hand has higher strength which may skew side effect reporting of weakness).

The evaluation of sweat production will be done using the subjective patient reported Hyperhidrosis Disease Severity Scale (HDSS) and objective gravimetric measurement. Hyperhidrosis Disease Severity Scale (HDSS) is a scale from 1 to 4. Values of 1 or 2 represent Mild/moderate disease, and 3 or 4 represent severe disease. Successful treatment is indicated by improvement from 3 or 4 to 1 or 2. One point improvement in HDSS score is associated with 50% reduction in sweat production and a two-point improvement with an 80% reduction, according to the Canadian Hyperhidrosis Advisory Committee.

Gravimetric measurement includes collecting sweat secretion on standardized filter. Prior to any measurements, the subject will be asked to sit in a climate-controlled room for 15 min to allow for acclimatization. Filter paper is first weighed on a high-precision laboratory scale. The filter papers are then placed in the subject's palms for 5 minutes, and weighed again. This technique has already been used in other studies of hyperhidrosis [5]. The difference in the weight (g) will allow calculation of sweat secretion in grams per 5 minutes.

The subject's palm will be cleansed with gauze. Then the microneedle pretreatment will be performed on both palms. This will consist of rolling the microneedles into the skin for several seconds on the sides of the palm. The microneedles are solid and are long enough to penetrate the stratum corneum and enter the epidermis. Microneedles that are less than 700 micrometers in length have been shown to induce minimal pain, and our ongoing work with microneedles that were 650 micrometers in length was rated a 1 out of 10 on a visual analog pain scale (results of IRB# 282150). For this study, subjects will rate pain on a visual analog scale after the microneedle pretreatment as well.

Next a VapoMeter will be used to measure the water evaporation gradient on the skin. The Vapometer measures the transepidermal water loss (TEWL) and evaporation rates. Measurements will be performed with non-invasive devices that have been widely used for the study of skin barrier function (Figure 1) [6]. Each device has a flat-top chamber (approximate diameter of 1cm) that will come in contact with the skin surface during measurements. This device has a humidity sensor and does not deliver any energy into the skin. The subjects will not experience discomfort during and after the measurements. The electrode tip will be cleaned with alcohol wipes between subjects.

Next, the subject will asked to grade their discomfort with the pretreatment step on a 10 cm visual analog pain scale.

Next, botulinum toxin A solution will be mixed per standard protocol in the dermatology clinic and will be applied and evenly spread over the palm that was randomized for treatment with botulinum toxin A. The other palm will be treated with a placebo (saline). This will be followed by occlusion with an occlusive wrap such as saran wrap, a silicone based gel, or glove. The subject will be asked to keep the saran wrap, silicone gel, or glove in place for 1 hour. Botulinum toxin A is an FDA approved product for the treatment of hyperhidrosis.

Follow-up visits will be at 4-6 weeks post treatment. During the follow-up visit the patient will be asked about side effects or any adverse events. Also a repeat evaluation of sweat production will be done using the subjective patient reported Hyperhidrosis Disease Severity Scale (HDSS) and objective gravimetric measurement. They will also complete a global satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age and older (split-hand microneedle group only)
* 18 years of age and older (split-hand botulinum toxin A group)
* Subjects with palmar hyperhidrosis
* Do not meet any of the exclusion criteria

Exclusion Criteria:

* Subjects who smoke
* Subjects who have established allergy to topical botulinum toxin
* Subjects with a personal or family history of neuromuscular disorder
* Subjects who have had botulinum toxin to the hands in the past 6 months
* Subjects who have had other systemic anticholinergic therapy in the past 2 weeks
* Subjects with known thyroid related disorders or systemic infection.
* Subjects who are pregnant or who plan to become pregnant

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08-02 (Actual); Study Completion 2016-08-02 (Actual)

PRIMARY OUTCOMES:
subjective patient reported Hyperhidrosis Disease Severity Scale (HDSS) | 1 month follow up
  a scale from 1 to 4. Values of 1 or 2 represent Mild/moderate disease, and 3 or 4 represent severe disease.
objective gravimetric measurement | 1 month follow up
  collecting sweat secretion on standardized filter, difference in the weight (g) will allow calculation of sweat secretion in grams per 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- [Background] Sivamani RK, Stoeber B, Liepmann D, Maibach HI. Microneedle penetration and injection past the stratum corneum in humans. J Dermatolog Treat. 2009;20(3):156-9. doi: 10.1080/09546630802512679. PMID 19016065
- [Background] Sivamani RK, Liepmann D, Maibach HI. Microneedles and transdermal applications. Expert Opin Drug Deliv. 2007 Jan;4(1):19-25. doi: 10.1517/17425247.4.1.19. PMID 17184159
- [Background] Sivamani RK, Stoeber B, Wu GC, Zhai H, Liepmann D, Maibach H. Clinical microneedle injection of methyl nicotinate: stratum corneum penetration. Skin Res Technol. 2005 May;11(2):152-6. doi: 10.1111/j.1600-0846.2005.00107.x. PMID 15807814